CLINICAL TRIAL: NCT06228989
Title: Restoration or Extraction as Dental Therapy in First Permanent Molars With Severe Hypomineralized Enamel (MIH) - a National Randomized Prospective Multicenter Study
Brief Title: Analysis of Treatment Outcomes in Patients Affected by Molar-Incisor Hypomineralization (MIH)
Acronym: GuREx-MIH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Region Östergötland (Other); Malmö University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 276481
Record Dates: First submitted 2024-01-03; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Hypomineralization of Enamel; Dental Fear; Quality of Life
MeSH Terms: conditions — Dental Enamel Hypomineralization

STUDY DESIGN:
Intervention Model Description: A multicentre prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Extraction therapy (Experimental): Patients exclusive treated with extraction therapy of any first permanent molars due to severe MIH.
  Affected first permanent molars were dignosed with MIH degree 4-6.
  Interventions: Procedure: Extraction therapy
- Restorative therapy (Experimental): Patients exclusive treated with restorative therapy of any first permanent molars due to severe MIH.
  Affected first permanent molars were dignosed with MIH degree 4-5.
  Interventions: Procedure: Restorative therapy
- Extraction therapy and Restorative therapy (Experimental): Patients undergoing combined treatment of both extraction therapy and restorative therapy of their first permanent molars due to MIH.
  Affected first permanent molars treated with extraction therapy were dignosed with MIH degree 6.
  Affected first permanent molars treated with restorative therapy were dignosed with MIH degree 4-5.
  Interventions: Procedure: Restorative therapy; Procedure: Extraction therapy
- Control patients (No Intervention): Patients devoid of any enamel developmental defects, attending the Public Dental Service in Region Västra Götaland, constituted a basis for the control patients. These controls were matched in terms of gender, age, and socio-economic factors, with each study patient paired with seven potential control patients.

INTERVENTIONS:
Procedure: Restorative therapy — Restorative treatment of first permanent molars affected with severe MIH
  Arms: Extraction therapy and Restorative therapy; Restorative therapy
Procedure: Extraction therapy — Extraction treatment of first permanent molars affected with severe MIH
  Arms: Extraction therapy; Extraction therapy and Restorative therapy

SUMMARY:
The aim is to long-term evaluate extraction or restoration therapy, of first permanent molars with extensive treatment needs as a result of severe MIH in a national multicenter study concerning dental fear and anxiety, oral health-related quality of life, jaw development, and health economics.

DETAILED DESCRIPTION:
First permanent molars often show areas of porous and hypomineralized enamel. This manifests itself clinically as whitish-yellow to brownish well-defined spots and, in severe disorders, disintegration of enamel. One to all molars are affected and at the same time, the permanent incisors may show opacities. The condition is called Molar-Incisor Hypomineralization (MIH) and occurs in 14% of children globally.

Affected teeth create problems for the individual. The teeth are often painful, e.g. when brushing teeth, cold food/drink, or even when inhaling cold air. Dental treatment can be painful because it is difficult to get adequate anesthesia, probably due to subclinical pulp inflammation caused by the porosity of the enamel.

Molars with severely demineralized enamel need dental care shortly after they have erupted due to decay and subsequent caries. 9-year-old children with severe MIH had their PFM treated almost ten times as often as a healthy control group. In case of widespread decay and hypersensitivity, extraction may be a treatment option.

Two retrospective studies dealing with the extraction of first permanent molars due to MIH have been published: one study found that 87% showed acceptable gap closure and another study showed that 3 of 27 extraction cases had an objective need and only one case had a subjective need for orthodontic gap closure after the extraction. A review article discusses the scientific basis for treating severe first permanent molar due to severe MIH, and the author claims that both the profession and the public today believe in a more conservative restorative treatment. However, he states that there is a need for well-controlled long-term studies.

The aim is to long-term evaluate extraction or restoration therapy, of first permanent molars with extensive treatment needs as a result of severe MIH in a national multicenter study concerning dental fear and anxiety, oral health-related quality of life, jaw development, and health economics.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-9 years
* Diagnosed with at least one first permanent molar with MIH defree 4-6

Exclusion Criteria:

* Dental agenesis
* General disorders, including chronic diseases and functional limitations

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2028-09-04 (Estimated)

PRIMARY OUTCOMES:
Dental fear and anxiety | At baseline - age 6-9 years (T0), At 1st follow-up - age 11 years (T1), At 2nd follow-up - age 15 years (T2))
  Questionnaire: Children's Fear Survey Schedule - Dental Subscale (CFSS-DS). Range 15-75, lower score indicated lower dental fear and anxiety
Oral helth-related quality of life | At baseline - age 6-9 years (T0), At 1st follow-up - age 11 years (T1), At 2nd follow-up - age 15 years (T2))
  Questionnaire: Short form of Child Perceptions Questionnaire for 11-14-year-old children (CPQ11-14).
  Range 0-64, lower score indicated better oral helth-related quality of life
Health economics | At baseline - age 6-9 years (T0), At 1st follow-up - age 11 years (T1), At 2nd follow-up - age 15 years (T2))
  Journal extract: nummber of dental visits and the length of dental visits. More dental chairtime indicates a higher health economic impact.

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Robertson, Principal Investigator — Göteborg University

IPD SHARING:
Plan to Share IPD: Yes
As soon as we finish with the data collection and the manuscript writing, the data will be published online.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After 2028
Access Criteria: The data will be de-identified